CLINICAL TRIAL: NCT04541810
Title: Post-marketing Surveillance to Evaluate the Safety and Effectiveness of Upadacitinib in Korean Patients
Brief Title: A Study of Oral Upadacitinib (RINVOQ) Tablets to Assess Adverse Events and Change in Disease Symptoms in Korean Participants With Moderate to Severe Active Rheumatoid Arthritis, Atopic Dermatitis, Ankylosing Spondylitis or Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-319
Record Dates: First submitted 2020-08-31; First posted 2020-09-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Rheumatoid Arthritis (RA); Atopic Dermatitis (AD); Ankylosing Spondylitis (AS); Psoriatic Arthritis (PsA)
Keywords: Rheumatoid Arthritis; Atopic Dermatitis (AD); Ankylosing Spondylitis (AS); Psoriatic Arthritis (PsA); Upadacitinib; RINVOQ
MeSH Terms: conditions — Arthritis, Rheumatoid; Dermatitis, Atopic; Spondylitis, Ankylosing; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants receiving Upadacitinib: Participants receiving Upadacitinib as prescribed by their physician per local label.

SUMMARY:
Rheumatoid Arthritis (RA) is an inflammatory disease of the joints characterized by the swelling of multiple joints and tenderness caused by progressive inflammatory synovitis, which leads to serious and debilitating diseases. Atopic dermatitis (AD) is a skin condition that may cause a rash and itching due to inflammation of the skin. Ankylosing Spondylitis (AS) is a form of chronic arthritis causing inflammation in the spine. This can cause pain and stiffness in the back. Psoriatic arthritis (PsA) is a type of arthritis (swelling and stiffness in the joints) that is frequently seen in trial participants who also have the skin condition psoriasis. It is caused by the body's immune system mistakenly attacking healthy joint tissue causing inflammation, joint damage, disability, and a reduced life expectancy. This study will assess the adverse events and change in disease symptoms in Korean participants with RA, AD, AS or PsA.

Upadacitinib is a drug approved for the treatment of moderately to severely active rheumatoid arthritis, atopic dermatitis, ankylosing spondylitis or psoriatic arthritis. Korean participants who have been prescribed upadacitinib by their physicians will be enrolled. Approximately, 3600 participants will be enrolled this study, in multiple sites within Korea.

Participants will receive Upadacitinib as prescribed by the physician and will be followed for approximately 28 weeks.

There will be no additional burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic and will be asked to provide additional information by questionnaire at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (>= 19 years of age), Atopic dermatitis includes both adolescents (>= 12 years of age) and adults.
* Participants suitable for the treatment with upadacitinib according to the approved local label.

Exclusion Criteria:

- Participants for whom the drug is contraindicated in the approved local label.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants receiving Upadacitinib according to the product prescribing information, for moderate to severe active Rheumatoid Arthritis (RA), Atopic Dermatitis (AD), Ankylosing Spondylitis (AS) or Psoriatic Arthritis (PsA).
Sampling Method: Non-Probability Sample
Enrollment: 2369 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | Up to approximately 6 years
  An adverse event (AE) is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with their treatment.
Percentage of Participants Achieving Responder Status Based on Disease Activity Score 28 Joints (DAS28) (Rheumatoid Arthritis Participants Only) | Up to 24 weeks
  Responder is a participant whose DAS28 at week 24 decreased by 1.2 or more compared to baseline.
Percentage of Participants Achieving Responder Status Based on Eczema Area and Severity Index (EASI) (Atopic Dermatitis Participants Only) | Up to 16 weeks
  Responder is a participant who achieve EASI 75.
Percentage of Participants Achieving Responder Status Based on Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) (Ankylosing Spondylitis Participants Only) | Up to 12 weeks
  Responder is a participant whose BASDAI at week 12 decreased by 50% or more than 2 compared to the baseline.
Percentage of Participants Achieving the Responder status Based on Active Joint Count (Psoriatic Arthritis Participants Only) | Up to 12 weeks
  Responder is a participant who achieve 30% or more reduction in Tender Joint Count and Swollen Joint Count compared to Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (116):
- South Korea (116):
  - Inje University - Busan Paik Hospital /ID# 259143, Busan, Busan Gwang Yeogsi
  - Haeundae Bumin Hospital /ID# 238959, Busan, Busan Gwang Yeogsi
  - Inje University Haeundae Hospital /ID# 238949, Busan, Busan Gwang Yeogsi
  - Dong-A University Medical Center /ID# 269937, Busan, Busan Gwang Yeogsi
  - Pusan National University Hospital /ID# 251315, Busan, Busan Gwang Yeogsi
  - Kosin University Gospel Hospital /ID# 239001, Busan, Busan Gwang Yeogsi
  - Dankook University Hospital /ID# 251307, Cheonan-si, Chungcheongnam-do
  - SoonChunHyang University Hospital Cheonan /ID# 248379, Cheonan-si, Chungcheongnam-do
  - SoonChunHyang University Hospital Cheonan /ID# 251302, Cheonan-si, Chungcheongnam-do
  - Kyungpook National University Hospital /ID# 251294, Daegu, Daegu Gwang Yeogsi
  - Kyungpook National University Hospital /ID# 251305, Daegu, Daegu Gwang Yeogsi
  - Chungnam National University Hospital /ID# 239000, Daejeon, Daejeon Gwang Yeogsi
  - Chungnam National University Hospital /ID# 259097, Daejeon, Daejeon Gwang Yeogsi
  - Daejeon Eulji Medical Center, Eulji University /ID# 251292, Daejeon, Daejeon Gwang Yeogsi
  - Daejeon Eulji Medical Center, Eulji University /ID# 251293, Daejeon, Daejeon Gwang Yeogsi
  - Konyang University Hospital /ID# 238951, Daejeon, Daejeon Gwang Yeogsi
  - Kangwon National University Hospital /ID# 248376, Chuncheon, Gang Weondo
  - Kangwon National University Hospital /ID# 259124, Chuncheon, Gang Weondo
  - Yonsei University-Wonju Severance Christian Hospital /ID# 239004, Wŏnju, Gang Weondo
  - Yonsei University-Wonju Severance Christian Hospital /ID# 239005, Wŏnju, Gang Weondo
  - Korea University Ansan Hospital /ID# 238992, Ansan-si, Gyeonggido
  - Korea University Ansan Hospital /ID# 251304, Ansan-si, Gyeonggido
  - Soon Chun Hyang University Hospital Bucheon /ID# 240935, Bucheon-si, Gyeonggido
  - Soon Chun Hyang University Hospital Bucheon /ID# 251321, Bucheon-si, Gyeonggido
  - The Catholic University Of Korea, Bucheon St. Mary'S Hospital /ID# 270022, Bucheon-si, Gyeonggido
  - The Catholic University of Korea, Bucheon St.Mary's Hospital /ID# 259142, Bucheon-si, Gyeonggido
  - Inje University - Ilsan Paik Hospital /ID# 270021, Goyang, Gyeonggido
  - Hanyang University Guri Hospital /ID# 259173, Guri-si, Gyeonggido
  - Hanyang University Guri Hospital /ID# 259175, Guri-si, Gyeonggido
  - Chung-Ang University Gwangmyeong Hospital /Id# 259180, Gwangmyeong, Gyeonggido
  - Chung-Ang University Gwangmyeong Hospital /ID# 270825, Gwangmyeong, Gyeonggido
  - Hallym University Dongtan Sacred Heart Hospital /ID# 259177, Hwaseong, Gyeonggido
  - Gachon University Gil Medical Center /ID# 262757, Incheon, Gyeonggido
  - Catholic Kwandong University International St.Mary's Hospital /ID# 248380, Incheon, Gyeonggido
  - CHA Bundang Medical Center /ID# 251324, Seongnam, Gyeonggido
  - CHA Bundang Medical Center /ID# 267001, Seongnam, Gyeonggido
  - Bundang Jesaeng Hospital /ID# 238999, Seongnam, Gyeonggido
  - Seoul National University Bundang Hospital /ID# 248378, Seongnam-si, Gyeonggido
  - Seoul National University Bundang Hospital /ID# 259115, Seongnam-si, Gyeonggido
  - Hallym University Sacred Heart Hospital /ID# 259150, Seoul, Gyeonggido
  - The Catholic University Of Korea St. Vincent's Hospital /ID# 245207, Suwon, Gyeonggido
  - The Catholic University Of Korea St. Vincent's Hospital /ID# 259149, Suwon, Gyeonggido
  - Ajou University Hospital /ID# 243488, Suwon, Gyeonggido
  - Ajou University Hospital /ID# 244494, Suwon, Gyeonggido
  - Ajou University Hospital /ID# 259123, Suwon, Gyeonggido
  - Uijeongbu Eulji Medical Center - Eulji University /ID# 259144, Uijeongbu-si, Gyeonggido
  - Uijeongbu Eulji Medical Center - Eulji University /ID# 270781, Uijeongbu-si, Gyeonggido
  - The Catholic University of Korea, Uijeongbu ST. Mary's Hospital /ID# 259182, Uijeongbu-si, Gyeonggido
  - Yongin Severance Hospital /ID# 238948, Yŏngin, Gyeonggido
  - Yongin Severance Hospital /ID# 251311, Yŏngin, Gyeonggido
  - Daegu Catholic University Medical Center /ID# 238996, Daegu, Gyeongsangbuk-do
  - Keimyung University Dongsan Hospital /ID# 259172, Daegu, Gyeongsangbuk-do
  - Keimyung University Dongsan Hospital /ID# 269942, Daegu, Gyeongsangbuk-do
  - Samsung Changwon Hospital /ID# 239003, Changwon, Gyeongsangnam-do
  - Changwon Fatima Hospital /ID# 238958, Changwon-si, Gyeongsangnam-do
  - Gyeongsang National University Changwon Hospital /ID# 269931, Changwon-si, Gyeongsangnam-do
  - Gyeongsang National University Hospital /ID# 267003, Jinju, Gyeongsangnam-do
  - Pusan National University Yangsan Hospital /ID# 239002, Yangsan, Gyeongsangnam-do
  - Pusan National University Yangsan Hospital /ID# 259120, Yangsan, Gyeongsangnam-do
  - The Catholic University of Korea, Incheon St. Mary's Hospital /ID# 240934, Incheon, Incheon Gwang Yeogsi
  - The Catholic University of Korea, Incheon St. Mary's Hospital /ID# 251306, Incheon, Incheon Gwang Yeogsi
  - The Catholic University of Korea, Incheon St. Mary's Hospital /ID# 269811, Incheon, Incheon Gwang Yeogsi
  - Inha University Hospital /ID# 251317, Incheon, Incheon Gwang Yeogsi
  - Design Hospital /ID# 262327, Jeollabuk-do, Jeonrabugdo
  - Jeonbuk National University Hospital /ID# 259140, Jeonju, Jeonrabugdo
  - Chosun University Hospital /ID# 259119, Gwangju, Jeonranamdo
  - Chonnam National University Hospital /ID# 251326, Gwangju, Jeonranamdo
  - Chungbuk National University Hospital /ID# 238997, Cheongju-si, North Chungcheong
  - Chungbuk National University Hospital /ID# 262334, Cheongju-si, North Chungcheong
  - Dr. Park's Internal Medicine Clinic /ID# 238995, Chungbuk, North Chungcheong
  - Konkuk University Chungju Hospital /ID# 240936, Chungju, North Chungcheong
  - Sejong Chungnam National University Hospital /ID# 238952, Sejong-si, Sejong-si
  - Sejong Chungnam National University Hospital /ID# 259216, Sejong-si, Sejong-si
  - Chungang University Hospital /ID# 238993, Dongjak-gu, Seoul Teugbyeolsi
  - Chungang University Hospital /ID# 251322, Dongjak-gu, Seoul Teugbyeolsi
  - Inje University Sanggye Paik Hospital /ID# 251316, Seoul, Seoul Teugbyeolsi
  - Nowon Eulji Medical Center, Eulji University /ID# 259139, Seoul, Seoul Teugbyeolsi
  - Seoul Medical Center /ID# 251310, Seoul, Seoul Teugbyeolsi
  - Kyung Hee University Hospital /ID# 259117, Seoul, Seoul Teugbyeolsi
  - Kyung Hee University Hospital /ID# 270182, Seoul, Seoul Teugbyeolsi
  - Korea University Anam Hospital /ID# 262333, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 245209, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 251319, Seoul, Seoul Teugbyeolsi
  - Kangbuk Samsung Hospital /ID# 238955, Seoul, Seoul Teugbyeolsi
  - Kangbuk Samsung Hospital /ID# 251308, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 259178, Seoul, Seoul Teugbyeolsi
  - SoonChunHyang University Seoul Hospital /ID# 259179, Seoul, Seoul Teugbyeolsi
  - SoonChunHyang University Seoul Hospital /ID# 269940, Seoul, Seoul Teugbyeolsi
  - National Medical Center /ID# 251303, Seoul, Seoul Teugbyeolsi
  - Hanyang University Seoul Hospital /ID# 238640, Seoul, Seoul Teugbyeolsi
  - Hanyang University Seoul Hospital /ID# 251320, Seoul, Seoul Teugbyeolsi
  - Konkuk University Medical Center /ID# 245208, Seoul, Seoul Teugbyeolsi
  - Rheuma Internal Clinic /ID# 238998, Seoul, Seoul Teugbyeolsi
  - Asan Bone Internal Medicine /ID# 238991, Seoul, Seoul Teugbyeolsi
  - Kyung Hee University Hospital at Gangdong /ID# 267000, Seoul, Seoul Teugbyeolsi
  - Kyung Hee University Hospital at Gangdong /ID# 267004, Seoul, Seoul Teugbyeolsi
  - VHS(Veterans Health Service) Medical Center /ID# 251323, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 251312, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital /ID# 270030, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 259152, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 245206, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 251314, Seoul, Seoul Teugbyeolsi
  - SMG-SNU Boramae Medical Center /ID# 238957, Seoul, Seoul Teugbyeolsi
  - SMG-SNU Boramae Medical Center /ID# 251325, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Yeouido ST. Mary's Hospital /ID# 251309, Seoul, Seoul Teugbyeolsi
  - Hallym University Kangnam Sacred Heart Hospital /ID# 262328, Seoul, Seoul Teugbyeolsi
  - Hallym University Kangnam Sacred Heart Hospital /ID# 270775, Seoul, Seoul Teugbyeolsi
  - Ewha Womans University Seoul Hospital /ID# 251327, Seoul, Seoul Teugbyeolsi
  - Ewha Womans University Medical Centre /ID# 270025, Seoul, Seoul Teugbyeolsi
  - Korea University Guro Hospital /ID# 259141, Seoul, Seoul Teugbyeolsi
  - HoYounKim's Clinic for Arthritis Rheumatism /ID# 238956, Seoul, Seoul Teugbyeolsi
  - Myungji Hospital /Id# 259148, Goyang
  - Yonsei University Health System Severance Hospital /ID# 248377, Seoul
  - Duplicate_Inje University Seoul Paik Hospital /ID# 238994, Seoul
  - Hallym University Kangdong Sacred Heart Hospital /ID# 251328, Seoul
  - Hallym University Sacred Heart Hospital /ID# 269934, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info. — https://www.abbvieclinicaltrials.com/study/?id=P20-319